CLINICAL TRIAL: NCT06952309
Title: Effect of Intravenous Lidocaine Combined With Intratracheal Dexmedetomidine on Postoperative Throat Pain in Patients Undergoing Thyroid Cancer Surgery
Brief Title: Intravenous Lidocaine Plus Intratracheal Dexmedetomidine on Postoperative Sore Throat
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anqing Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Xuwen531
Record Dates: First submitted 2025-04-20; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Dexmedetomidine; Lidocaine; Sore Throat
Keywords: dexmedetomidine; lidocaine; thyroid surgery; sore throat
MeSH Terms: conditions — Pharyngitis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intravenous lidocaine (Experimental): Group L received lidocaine 1.5 mg/kg was injected intravenously 3 min before endotracheal intubation and tracheal spray with 0.8% ropivacaine 40 mg (5 mL) for surface anesthesia
  Interventions: Drug: Intravenous lidocaine
- Intracheal dexmedetomidine (Experimental): Group D received equal volume normal saline was injected intravenously 3 min before tracheal intubation and tracheal spray with dexmedetomidine (1 μg/kg) mixed with 0.8% ropivacaine 40 mg (5 mL) for surface anesthesia
  Interventions: Drug: Intracheal dexmedetomidine
- Intravenous lidocaine combined with intracheal dexmedetomidine (Experimental): Group LD received lidocaine 1.5 mg/kg was injected intravenously 3 min before endotracheal intubation and tracheal spray with dexmedetomidine (1 μg/kg) mixed with 0.8% ropivacaine 40 mg (5 mL) for surface anesthesia
  Interventions: Drug: Intravenous lidocaine combined with intracheal dexmedetomidine
- Saline (Experimental): Group C received equal volume normal saline was injected intravenously 3 min before tracheal intubation and tracheal spray with 0.8% ropivacaine 40 mg (5 mL) for surface anesthesia
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: Intracheal dexmedetomidine — Group D received equal volume normal saline was injected intravenously 3 min before tracheal intubation and tracheal spray with dexmedetomidine (1 μg/kg) mixed with 0.8% ropivacaine 40 mg (5 mL) for surface anesthesia
  Arms: Intracheal dexmedetomidine
Drug: Intravenous lidocaine — Group L received lidocaine 1.5 mg/kg was injected intravenously 3 min before endotracheal intubation and tracheal spray with 0.8% ropivacaine 40 mg (5 mL) for surface anesthesia
  Arms: Intravenous lidocaine
Drug: Intravenous lidocaine combined with intracheal dexmedetomidine — Group LD received lidocaine 1.5 mg/kg was injected intravenously 3 min before endotracheal intubation and tracheal spray with dexmedetomidine (1 μg/kg) mixed with 0.8% ropivacaine 40 mg (5 mL) for surface anesthesia
  Arms: Intravenous lidocaine combined with intracheal dexmedetomidine
Drug: Saline (NaCl 0,9 %) (placebo) — Group C received equal volume normal saline was injected intravenously 3 min before tracheal intubation and tracheal spray with 0.8% ropivacaine 40 mg (5 mL) for surface anesthesia
  Arms: Saline

SUMMARY:
Objective: The present study was to investigate the effect of intravenous lidocaine combined with intratracheal dexmedetomidine on postoperative sore throat in patients undergoing thyroid cancer surgery.

Methods: Investigators enrolled 144 patients with American Society of Anesthesiologists (ASA) physical status I and II, aged 18-65 years, and scheduled for elective undergoing thyroid cancer surgery with general anesthesia. The participants were randomly assigned into four groups(n=36 each group): Group L received lidocaine 1.5 mg/kg was injected intravenously 3 min before endotracheal intubation and tracheal spray with 0.8% ropivacaine 40 mg (5 mL) for surface anesthesia. Group D received equal volume normal saline was injected intravenously 3 min before tracheal intubation and tracheal spray with dexmedetomidine (1 μg/kg) mixed with 0.8% ropivacaine 40 mg (5 mL). Group LD received lidocaine 1.5 mg/kg was injected intravenously 3 min before endotracheal intubation and tracheal spray with dexmedetomidine (1 μg/kg) mixed with 0.8% ropivacaine 40 mg (5 mL). Group C received equal volume normal saline was injected intravenously 3 min before tracheal intubation and tracheal spray with 0.8% ropivacaine 40 mg (5 mL) for surface anesthesia.The incidence and severity of postoperative sore throat were recorded in four groups at 1 h, 2 h, 6 h, 24 h and 48 h after operation.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid cancer surgery with ASA grades I-II
* Aged 18-65 years
* The patient's communication is normal and they have a certain learning ability

Exclusion Criteria:

* Severe respiratory and circulatory system diseases
* There was bradycardia (HR < 60 beats/minute) or atrioventricular block before the operation
* Nervous system disease
* Mental and psychological disorders
* Abnormal liver and kidney functions
* Pregnant and lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of postoperative sore throat | at 1 hour, 2 hour, 6 hour, 24 hour and 48 hour after operation

IPD SHARING:
Plan to Share IPD: No